CLINICAL TRIAL: NCT04565600
Title: Prevention of Taxane-associated Acute Pain Syndrome With Etoricoxib for Breast Cancer Patients: A Phase II Randomized Trial
Brief Title: Prevention of Taxane-associated Acute Pain Syndrome With Etoricoxib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20190516
Record Dates: First submitted 2020-09-13; First posted 2020-09-25 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Pain Syndrome
Keywords: Breast Cancer; Docetaxel; Etoricoxib; Acute pain syndrome; Peripheral neuropathy
MeSH Terms: conditions — Somatoform Disorders; Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoricoxib (Experimental): Prophylactic etoricoxib (60 mg) was administered orally at each course of docetaxel-containing chemotherapy, which started from the day of chemotherapy and was performed once per day for 8 days (day 1-8).
  Interventions: Drug: Etoricoxib
- Control (No Intervention): No prophylactic regimen was given.

INTERVENTIONS:
Drug: Etoricoxib — Etoricoxib 60 Mg Oral Tablet
  Arms: Etoricoxib

SUMMARY:
A phase II randomized clinical trial was conducted to determine whether etoricoxib could prevent or ameliorate the incidence and/or severity of docetaxel-induced acute pain syndrome. We also aimed to determine if there are any improvement of the late-onset peripheral neuropathy as well as quality of life with prophylactic etoricoxib for breast cancer patients who receive docetaxel chemotherapy.

DETAILED DESCRIPTION:
Docetaxel plays a key role in reducing the recurrence of early-stage breast cancer as well as improving survival outcomes of advanced breast cancer patients, but it causes a variety of adverse events, including myalgia and arthralgia, peripheral neuropathy, febrile neutropenia, and hypersensitivity reactions and so on. The myalgia and arthralgia induced by docetaxel, which have been together referred to as taxane-associated acute pain syndrome (T-APS), were reported to occur in 3.6% to 70% of patients, and the symptoms usually occurred 24-48 hours after docetaxel infusion and lasted for 3-5 days. Previous studies found that patients who experienced myalgia and arthralgia due to docetaxel administration were more likely to have chronic peripheral neuropathy, which supported that T-APS could be a form of neurologic toxicity. T-APS may significantly influence patients' sleep and daily life, and even caused discontinuation of chemotherapy. Therefore, it is clinically meaningful to explore some prophylactic drugs for the T-APS. Previous studies had used glutamine, corticosteroids, Shakuyaku-Kanzo-To (a Japanese herb), and gabapentin to prevent paclitaxel-induced myalgia and arthralgia, but failed to provide enough evidence for clinical practice. Etoricoxib, a selective COX-2 inhibitor, is a nonsteroidal anti-inflammatory drug (NSAID) that has showed comparable efficacy in acute and chronic pain, with fewer gastrointestinal (GI) adverse events compared with traditional NSAIDs. Therefore, we conducted a phase II randomized clinical trial to investigate whether etoricoxib could prevent or ameliorate the incidence and/or severity of docetaxel-induced acute pain syndrome. We also aimed to determine if there are any improvement of the late-onset peripheral neuropathy as well as quality of life with prophylactic etoricoxib for breast cancer patients who receive docetaxel chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18 years
* Stage I-III breast cancer
* ECOG 0-2
* Received docetaxel-containing chemotherapy

Exclusion Criteria:

* Existed any chronic pain or peripheral neuropathy
* Prior history of gastrointestinal bleeding or ulcer
* Long-term history of receiving oral corticoids, nonsteroid anti-inflammatory drugs (NSAIDs) or anti-histamines
* Allergies to NSAIDs or aspirin
* Blood creatinine level exceeds 1.5 times of the upper limit of normal range

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
overall incidence of taxane-associated acute pain syndrome across all cycles of chemotherapy | 6 months
  Total incidence of myalgia and arthralgia of patients across all cycles of docetaxel chemotherapy

SECONDARY OUTCOMES:
incidence of taxane-associated acute pain syndrome at each cycle | 6 months
  Incidence of myalgia and arthralgia of patients at each cycle of docetaxel chemotherapy
severity of taxane-associated acute pain syndrome at each cycle | 6 months
  Severity of myalgia and arthralgia of patients at each cycle of docetaxel chemotherapy; the severity of pain was evaluated on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
duration of taxane-associated acute pain syndrome at each cycle | 6 months
  Duration of myalgia and arthralgia of patients at each cycle of docetaxel chemotherapy; the duration of pain was counted by days.
incidence of severe taxane-associated acute pain syndrome by cycle and across all cycles | 6 months
  incidence of severe myalgia and arthralgia (score, defined as greater than 5 on a scale from 0 to 10) of patients during the period of docetaxel chemotherapy by cycle and across all cycles
Functional Assessment of Cancer Therapy-Breast (FACT-B) subscale at each cycle | 6 months
  Functional Assessment of Cancer Therapy-Breast（FACT-B）subscale during the period of docetaxel chemotherapy was assessed; the scores range from 0 to 144, higher scores mean a better outcome (higher quality of life)
incidence of peripheral neuropathy after all cycles of chemotherapy | 6 months
  Functional Assessment of Cancer Treatment Neurotoxicity (FACT-Ntx) subscale (FACT-Ntx score <44), Eastern Cooperative Oncology Group neuropathy scale (ENS) subscale and EMG were performed at 3 months after the completion of chemotherapy.
adverse events | 6 months
  Assessment of adverse events was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang J, Gao HF, Yang C, Zhu T, Ji F, Yang M, Zhang L, Li J, Cheng M, Zhang T, Shen B, Chen Y, Wang K. Prevention of taxane-associated acute pain syndrome with etoricoxib for patients with breast cancer: A phase II randomised trial. Eur J Cancer. 2022 Aug;171:150-160. doi: 10.1016/j.ejca.2022.05.019. Epub 2022 Jun 17. PMID 35724467